CLINICAL TRIAL: NCT03628430
Title: Effect of Buffered Lidocaine With Epinephrine in Local Anesthesia During Subcutaneous Implantable Venous Access Devices Insertion: Double Blind Randomized Study.
Brief Title: Effect of Buffered Lidocaine With Epinephrine in Local Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Mohamed Kahloul, principal investigator, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HFH2922016
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Pain; Anesthesia, Local
Keywords: Anesthesia;; lidocaine;; patient experience; patient pain; sodium bicarbonate; Vascular Access Devices
MeSH Terms: conditions — Pain | interventions — Lidocaine; Epinephrine; Sodium Bicarbonate; Saline Solution

STUDY DESIGN:
Intervention Model Description: participants were assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Placebo Comparator): For patients of this group, the intervention was a Local Anesthesia with:
  * 10 mL of 2% lidocaine with epinephrine 0.005mg/ml
  * and 5 mL of 0.9% NaCl
  Interventions: Procedure: lidocaine with epinephrine; Procedure: Normal saline
- Group A (Active Comparator): For patients of this group, the intervention was a Local Anesthesia with:
  * 10 mL of 2% lidocaine with epinephrine 0.005mg/ml
  * and 5 mL of 4.2 % sodium bicarbonate
  Interventions: Procedure: lidocaine with epinephrine; Procedure: sodium bicarbonate

INTERVENTIONS:
Procedure: lidocaine with epinephrine — Local anesthesia with lidocaine with epinephrine
Procedure: sodium bicarbonate — sodium bicarbonate as adjuvant to lidocaine with epinephrine in Local anesthesia
  Arms: Group A
Procedure: Normal saline — normal saline as adjuvant to lidocaine with epinephrine in Local anesthesia
  Arms: Group C

SUMMARY:
Subcutaneous implantable venous access devices are routinely implanted under local anesthesia. However, patients complain of pain during the injection of local anesthesia. The aim of this study was to evaluate the effectiveness of sodium bicarbonate-buffered lidocaine with epinephrine on reducing pain and patients' satisfaction during subcutaneous implantable venous access devices insertion.

A prospective double-blind study was conducted over a period of 6 months (1st January 2017 to 30th June 2017). Patients were randomized to receive either buffered (PH= 7.33) or plane lidocaine (PH= 3.50). The same operator made all insertions using a standard technique. Pain at five procedural steps (local anesthetic infiltration, central vein cannulation, skin incision, deep tissue dissection and pocket formation, and skin closure) and satisfaction were evaluated on a VAS score (0-100 mm). Secondary outcomes were sensory block onset time using pinprick test and patients' satisfaction.

DETAILED DESCRIPTION:
This prospective, randomized, controlled, double-blinded study was carried out in the Anesthesia and Resuscitation Department of Farhat Hached University Hospital of Sousse over a period of 6 months (1st January 2017 to 30th June 2017). Ethical approval was obtained from the institution's Research Ethics Board. Written informed consent was obtained from each patient by the investigators before entering this study. Outpatients, aged over 18 years, scheduled for Porta-Cath (PAC) insertion under local anesthesia were included.

Apart from the usual contraindications to PAC insertion, pregnant women, patients with a known allergy to study drugs, patients chronically using opioids or benzodiazepine for cancer or chronic pain, patients with history of thoracic or cervico-facial radiotherapy or those with severe cardiovascular and respiratory compromise or having a neuropathy were excluded from the study.

The study subjects randomly received, in a double blind manner (using computer-generated allocation numbers sealed in brown envelopes), one of two local anesthetic solutions. The pH adjusted group (group A) received 5 mL of 4.2 % sodium bicarbonate added to 10 mL of 2% lidocaine with epinephrine 0.005mg/ml (Lidocaine adrenaline; Aguettant, France) and the control group (group C) received 5 mL of 0.9% NaCl added to 10 mL of 2% lidocaine with epinephrine 0.005mg/ml (Lidocaine adrenaline; Aguettant, France).

Local anesthetic solutions were freshly prepared by a member of the anesthesia team and balanced at room temperature 30 minute prior to the procedure, whereas the anesthetist in charge of the patient was unaware of the prepared solution. The pH values of the final formulations have been measured using a pH-meter (PH-meter/millivoltmeter 3510 JENWAY) at the beginning of the study; it was 3.5 in the control group and 7.33 in the study group.

Routine monitoring included heart rate, blood pressure, oxyhemoglobin saturation, and respiratory rate were applied at arrival in the operating room. The process has been carried out in conditions of surgical asepsis. The preparation of the insertion area of the PAC included a prerequisite depilation, a cleaning of the area, rinsing, drying, an application of an antiseptic and then the setting of sterile drapes widely extending beyond the catheterization area. No preoperative sedation was administered. There was no pretreatment of the skin with any type of topical anesthetic or pain reducing technique before the injection of the anesthetic mixture.

The operator was provided with a syringe containing one of the randomly assigned local anesthetics. After confirming suitability of the target subclavian vein by ultrasound, the operator injected 3 mL of the local anesthetic solution through a 25 gauge needle directly superficial to the subclavian vein with ultrasound guidance. This injection was deliberate and not rushed, lasting 10 sec, with the same angle of injection with regard to the skin. The needle was then repositioned to inject 12mL to infiltrate the skin and deep tissue of the targeted area of the anterior chest wall. Each patient received a 7 Fr catheter via a non-tunneled approach. Each patient underwent instruction on rating pain and satisfaction via a standardized 100 mm horizontal linear visual analog scale (VAS) in which a score of 0 represented no pain / not satisfied and 100 represented the worst possible pain /very satisfied.

The primary outcome of this study was pain assessed on VAS at five procedural steps: 1) local anesthetic infiltration, 2) central vein cannulation, 3) skin incision, 4) deep tissue dissection and pocket formation, and 5) skin closure. Secondary outcomes were sensory block onset time using pinprick test and patients' satisfaction.

The required sample size was calculated hoping for a decrease of 30 mm of the VAS score during the injection of the local anesthetic after alkalinization, with a power (1-β) of 90%, a non-directional risk α of 5%, and assuming a standard deviation of 42, the size of the sample per group was estimated at 42. The sample size was increased to 60 patients per group in order to prevent the possible missing data or violation of the protocol.

Data were collected on customized data collection sheets and analyzed by the dedicated statistical software (IBM® Statistical Package for Social Science (SPSS), version 21.0, New York, USA). A p value of 0.05 was considered statistically significant. The quantitative variables were expressed in average and standard deviation. The qualitative variables were expressed in numbers and percentage. In order to compare qualitative variables, Pearson Chi-2 test was used. Student's t-test was used to compare quantitative variables.

ELIGIBILITY:
Inclusion Criteria:

Outpatients, aged over 18 years, scheduled for PAC placement under local anesthesia

Exclusion Criteria:

* usual contraindications to PAC insertion,
* pregnant women,
* patients with a known allergy to study drugs,
* patients chronically using opioids or benzodiazepine for cancer or chronic pain,
* patients with history of thoracic or cervico-facial radiotherapy
* patients with severe cardiovascular and respiratory compromise
* patients having a neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
T1 pain intensity | Immediately after local anesthetic infiltration
  pain intensity assessed immediately after local anesthetic infiltration, by a 100 mm visual analog scale (VAS) ranging from 0 (no pain) to 100 (the worst possible pain).
T2 pain intensity | Immediately after central vein cannulation
  pain intensity assessed immediately after central vein cannulation, by a 100 mm visual analog scale (VAS) ranging from 0 (no pain) to 100 (the worst possible pain).
T3 pain intensity | Immediately after skin incision,
  pain intensity assessed immediately after skin incision, by a 100 mm visual analog scale (VAS) ranging from 0 (no pain) to 100 (the worst possible pain).
T4 pain intensity | Immediately after deep tissue dissection and pocket formation,
  pain intensity assessed immediately after deep tissue dissection and pocket formation, by a 100 mm visual analog scale (VAS) ranging from 0 (no pain) to 100 (the worst possible pain).
T5 pain intensity | Immediately after skin closure.
  pain intensity assessed immediately after skin closure, by a 100 mm visual analog scale (VAS) ranging from 0 (no pain) to 100 (the worst possible pain).

SECONDARY OUTCOMES:
sensory block onset time | up to one hour after the intervention
  sensory block onset time assessed by pinprick test
patients' satisfaction. | Immediately after the intervention
  patients' satisfaction assessed by a 100 mm visual analog scale (VAS) ranging from 0 (not satisfied) to 100 (very satisfied).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kirk LM, Brown SD, Luu Y, Ogle A, Huffman J, Lewis PO. Beyond-use dating of lidocaine alone and in two "magic mouthwash" preparations. Am J Health Syst Pharm. 2017 May 1;74(9):e202-e210. doi: 10.2146/ajhp160214. PMID 28438825
- [Result] Phero JA, Nelson B, Davis B, Dunlop N, Phillips C, Reside G, Tikunov AP, White RP Jr. Buffered Versus Non-Buffered Lidocaine With Epinephrine for Mandibular Nerve Block: Clinical Outcomes. J Oral Maxillofac Surg. 2017 Apr;75(4):688-693. doi: 10.1016/j.joms.2016.09.055. Epub 2016 Oct 8. PMID 27815105
- [Result] Vasan A, Baker JA, Shelby RA, Soo MSC. Impact of Sodium Bicarbonate-Buffered Lidocaine on Patient Pain During Image-Guided Breast Biopsy. J Am Coll Radiol. 2017 Sep;14(9):1194-1201. doi: 10.1016/j.jacr.2017.03.026. Epub 2017 May 17. PMID 28527821
- [Result] Lee HJ, Cho YJ, Gong HS, Rhee SH, Park HS, Baek GH. The effect of buffered lidocaine in local anesthesia: a prospective, randomized, double-blind study. J Hand Surg Am. 2013 May;38(5):971-5. doi: 10.1016/j.jhsa.2013.02.016. Epub 2013 Apr 6. PMID 23566722
- [Result] Welch MN, Czyz CN, Kalwerisky K, Holck DE, Mihora LD. Double-blind, bilateral pain comparison with simultaneous injection of 2% lidocaine versus buffered 2% lidocaine for periocular anesthesia. Ophthalmology. 2012 Oct;119(10):2048-52. doi: 10.1016/j.ophtha.2012.05.029. Epub 2012 Jul 6. PMID 22771049